CLINICAL TRIAL: NCT06732180
Title: An Open-label Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GT-02287 in Participants With Parkinson's Disease With or Without a Pathogenic GBA1 Mutation
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GT-02287 in Parkinson's Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gain Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GANX-001-V102
Record Dates: First submitted 2024-12-09; First posted 2024-12-13 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single-arm. All participants receive the active molecule (once daily GT-02287 administration) (Experimental)
  Interventions: Drug: GT-02287

INTERVENTIONS:
Drug: GT-02287 — Dose of 13.5 mg/kg/day (plus/minus 2 mg/kg/day based on body weight) to be administered orally once a day for 90 days. Dosage form: powder in sachet (200 mg of GT-02287 per sachet) for reconstitution with a suspending agent

SUMMARY:
The main goal of this clinical trial is to learn about the safety and tolerability of GT-02287. The questions it aims to answer are:

* What medical problems do participants have when taking GT-02287?
* How is GT-02287 absorbed, distributed, and removed from the body of participants over time (pharmacokinetics)?
* Are there any biological effects of GT-02287 in blood and in cerebrospinal fluid that could be beneficial for people with Parkinson's disease?

Participants will:

* visit the clinic to assess if they qualify for the study (30-day Screening Period)
* if eligible, receive GT-02287 once a day every day for 90 days (90-day Open Label Treatment period)
* visit the clinic the first day of treatment, after the first 2 weeks of treatment, and every month during the 90-day Treatment Period.
* visit the clinic to assess how they are doing 14 days after the end of GT-02287 treatment (14-day Follow-Up Period).

DETAILED DESCRIPTION:
This Phase 1b, 3-month, multicenter, open-label study of GT-02287 in participants with Parkinson's Disease with or without GBA1 mutations. The primary objective of the study is to evaluate the safety and tolerability of GT-02287. The study will also investigate pharmacokinetics (PK) and explore pharmacodynamic parameters in blood and CSF and effect of GT-02287 on scores from selected clinical scales. Approximately 20 participants will be enrolled to result in approximately 15 evaluable participants.

All participants will receive an oral dose of GT-02287 of 13.5 mg/kg/day (plus/minus 2 mg/kg/day) once a day for 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent and be willing to comply with the requirements and restrictions of the study
* Any sex, ≥30 and ≤85 years of age
* Diagnosis of PD based on MDS criteria
* Within 7 years of PD diagnosis
* Body mass index of ≥18 and ≤40 kg/m2, and a body weight ≥45 kg and ≤120 kg
* Willing to provide a blood sample for PD-related genetic testing
* Hoehn & Yahr 1-3, inclusive
* No severe motor fluctuations or disabling dyskinesias based on the investigator's clinical assessment
* Naïve to pharmacological treatment for PD or on stable PD medication for ≥3 months prior to Screening, including ≥4 weeks at the same dose(s) immediately before Screening
* Not pregnant or breastfeeding
* If participant is either of childbearing potential or produces potentially viable sperm, participant must agree to use 2 forms of contraception (barrier method and a second highly effective form of birth control/contraception, as defined in the protocol) if engaging in potentially reproductive intercourse (with a partner who produces potentially viable sperm or is of childbearing potential, respectively)
* Agreeing to not participate in another investigational study while taking part in this study
* For participants with known GBA1 mutations, presence of a GBA1 mutation that has been associated with an increased risk of PD

Exclusion Criteria:

* Other neurological disorders, including but not limited to Alzheimer's disease, amyotrophic lateral sclerosis, frontotemporal dementia, progressive supranuclear palsy, corticobasal syndrome, Huntington's disease, multiple system atrophy, dementia with Lewy bodies, secondary (e.g. drug-induced) parkinsonism, multiple sclerosis, or epilepsy
* A history of Gaucher disease or homozygous for a GBA1 pathogenic variant known to be associated with GD or compound heterozygous for 2 alleles that are known to be associated with GD.
* Known PD-associated LRRK2 pathogenic variant or other PD-associated genetic mutations other than GBA1
* Dementia or a moderate cognitive impairment (score ≥17 on the Montreal Cognitive Assessment)
* Hypersensitivity to GT-02287 or any of its excipients
* Concomitant medications metabolized primarily by cytochrome P450 3A4 (CYP3A4) that have a narrow therapeutic window, concomitant medications that are substrates of breast cancer resistance protein and/or P-glycoprotein and that have a narrow therapeutic window, concomitant medications that are potent inhibitors or inducers of CYP3A4
* Use of dopamine antagonists (antipsychotics) or anticholinergic medications
* Concomitant disease including, but not limited to cardiovascular conditions, diabetes, autoimmune disease, cancer, active infectious disease, psychotic disorders and symptoms, depressive symptoms, drug and/or alcohol misuse as defined in the protocol
* Malabsorption or relevant disorder which may impact the absorption of GT-02287
* Clinically significant abnormalities in laboratory test
* Contraindications to lumbar puncture (LP)
* Blood donation >500 mL within 3 months
* Unable to comply with restrictions on food products, smoking, and /or alcohol use as defined in protocol
* participation in any interventional clinical study within 3 months or 5 half-lives, whichever is longer, prior to Screening

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence, nature, relationship to investigational product (IP), and severity of adverse events (AEs) | From first dose to Day 105
Incidence of clinically significant findings for clinical laboratory evaluations, physical and neurological examinations, body weight , vital signs measurements, 12-lead o 12-lead electrocardiograms (ECGs), Columbia Suicide Severity Rating Scale (C-SSRS) | From first dose to Day 105

SECONDARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | Day 1 and Day 90
  Pharmacokinetics
Area under the curve [AUC] | Day 1 and Day 90
  Pharmacokinetics
Time to reach Cmax [Tmax] | Day 1 and Day 90
  Pharmacokinetics
Elimination half life [T1/2] | Day 90- Day 93
  Pharmacokinetics
Apparent Clearance (CL/F) | Day 90- Day 93
  Pharmacokinetics
Apparent Volume of Distribution (Vz/F) | Day1 and Day 90- Day 93
  Pharmacokinetics

OTHER OUTCOMES:
Gcase activity (µmol/L/h) measurement in dried blood spots (DBS) | From first dose to Day 90
  Pharmacodynamics (Exploratory outcome): mean change from baseline in Gcase activity in DBS
Concentration of sphingolipids in cerebrospinal fluid (CSF ) | From first dose to Day 90
  Pharmacodynamics (Exploratory outcome): mean change from baseline in sphingolipids in CSF

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Gain Therapeutics, Inc.
Locations (7):
- Australia (7):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Southern Neurology, Kogarah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - CMAX, Adelaide, South Australia
  - Alfred Health, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: No